CLINICAL TRIAL: NCT05956444
Title: Effect of Neurodevelopmental Treatment on Fall Risk and Balance in Children With Spastic Cerebral Palsy
Brief Title: NDT on Fall Risk in Cerebral Palsied Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fatih Tekin, Assist. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FallRisk
Record Dates: First submitted 2023-07-06; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Palsy, Spastic; Falling
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Treated with both the treatment programs determined on the basis of the NDT and conventional physiotherapy. Programs prepared specifically for each child, in a 45-minute single session, 2 days a week, for 8 weeks in total. Each child was given a treatment program tailored to their needs.
  Interventions: Other: Neurodevelopmental Therapy (NDT); Other: Conventional Physiotherapy
- Control Group (Active Comparator): Treated with only the treatment programs determined on the basis of conventional physiotherapy.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Neurodevelopmental Therapy (NDT) — In the treatment program; vestibular and proprioceptive training on the balance board; dynamic balance training in sitting with eyes open and closed, kneeling upright and standing; balance exercises in front of the mirror; standing on one leg with eyes open and closed to increase proprioceptive input; vestibular and proprioceptive training on exercise balls of the appropriate size; balance training on the trampoline; footpad sensory stimulation with different materials; weight-bearing training in sitting, crawling, kneeling and standing positions; functional reaching and throwing-holding exercises in different positions; multitasking pieces of training; gait exercises in various ways and training for climbing and descending stairs appropriate to the child's situation (assisted, unaided, symmetrical, reciprocal) took place.
  Arms: Treatment Group
Other: Conventional Physiotherapy — Classical physiotherapy applications for balance.

SUMMARY:
Children with spastic cerebral palsy experience falls due to weakness in balance skills and abnormalities in gait parameters. It is necessary to improve the quality of life of these children by reducing the frequency of falling. Aim of this study was to investigate the effect of Neurodevelopmental Treatment on the risk of falling and balance and to contribute to the literature on this subject. Cases were randomized into study and control groups. At the beginning of the study, the balance skills of all the cases with spastic cerebral palsy were measured with the Pediatric Balance Scale, and the gait parameters and fall risks were measured with the LEGSys Temporospatial Gait Analysis Device. Then, an 8-week, case-specific, neurodevelopmental therapy program with intensive gait and balance training was applied to the study group in a 45-minute single session, 2 days a week. The control group received 8 weeks of conventional physiotherapy. At the end of the treatment process, the evaluations were repeated with the same methods.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy diagnosis
* Spastic type
* Gross Motor Function Classification System Level I and II

Exclusion Criteria:

* Tendon release surgery or Botox application in the last 6 months

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
LEGSys, Temporospatial Gait Analysis Device | Beginning of the study
  Determining the patient's risk of falling by performing a kinetic analysis of the gait
LEGSys, Temporospatial Gait Analysis Device | 8 weeks
  Determining the patient's risk of falling by performing a kinetic analysis of the gait
Pediatric Balance Scale (PBS) | Beginning of the study
  Functional balance was assessed using PBS, which consists of fourteen tasks similar to activities of daily living. Higher scores indicate better balance.
Pediatric Balance Scale (PBS) | 8 weeks
  Functional balance was assessed using PBS, which consists of fourteen tasks similar to activities of daily living. Higher scores indicate better balance.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Tekin, Prof., Study Chair — Faculty Member
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)